CLINICAL TRIAL: NCT05059717
Title: Imaging Tissue Motion Using MR Displacement Encoding With Stimulated Echo (DENSE): Detection of Early Chemotherapy Related Liver Injury Prior to Resection of Colorectal Liver Metastases
Brief Title: An Investigational Scan (MR DENSE) in Detecting Early Chemotherapy-Related Liver Injury Before Surgery in Patients With Resectable Colorectal Liver Metastases
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Overall Recruitment Status Withdrawn no participants
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-1115; NCI-2019-02483 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-1115 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-09-09; First posted 2021-09-28 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Colorectal Carcinoma Metastatic in the Liver
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (standard of care MRI, MR DENSE MRI) (Experimental): Patients undergo standard of care MRI and then undergo an MRI of the liver using MR DENSE imaging sequences over 60-90 minutes. Healthy volunteers undergo MRI of the liver using DENSE imaging sequences.
  Interventions: Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Procedure: Magnetic Resonance Imaging — Undergo standard of care MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Magnetic Resonance Imaging — Undergo MR DENSE imaging
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging

SUMMARY:
This trial studies how well a magnetic resonance imaging technique called Displacement Encoding with Stimulated Echo (DENSE) works in detecting chemotherapy-related liver injury in patients with colorectal cancer that has spread to the liver and can be removed by surgery. Researchers want to learn if the DENSE technique improves the standard MRI method.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. This is an exploratory study to collect Magnetic Resonance Displacement Encoding with Stimulated Echo (MR DENSE) imaging data of patients treated with chemotherapy prior to resection of metastases to explore its utility in detecting sinusoidal liver injury.

SECONDARY OBJECTIVES:

I. Estimate sensitivity of MR DENSE (determine degree of 2 dimensional [2D] vector displacement with cardiac cycle and variability of measurements with cardiac ventricle contraction).

II. Determine detection of sinusoidal injury (sinusoidal fibrosis, necrosis of pericentral hepatocytes, narrowing and fibrosis of central veins) on biopsy with non-alignment of 2D point vectors (horizontal and vertical direction) from neighboring/immediate adjacent points on MR DENSE imaging.

III. Determine correlation of intra-operative surgical scores (liver color and texture) with non-alignment of 2D point vectors (horizontal and vertical direction) from neighboring/immediate adjacent points on MR DENSE imaging.

OUTLINE:

Patients undergo standard of care magnetic resonance imaging (MRI) and then undergo an MRI of the liver using MR DENSE imaging sequences over 60-90 minutes. Healthy volunteers undergo MRI of the liver using DENSE imaging sequences.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with neoadjuvant chemotherapy and scheduled for hepatectomy, per standard of care at our institution, and meet criteria for hepatectomy.
* No contraindications to MRI (such implanted ferromagnetic or pump devices, metallic fragments in eye), as indicated on our departmental MRI screening form.
* Patient who is able to undergo informed consent.
* Men and non-pregnant women.
* Metastatic disease limited to liver.
* Metastases involving no more than 6 liver segments.
* No radiographic evidence of involvement of the hepatic artery, major bile ducts, main portal vein, celiac/para aortic lymph nodes.

Exclusion Criteria:

* Contraindication to MRI.
* Inability to comply with study and/or follow-up procedures.
* Unable to provide informed consent.
* Presence of extrahepatic metastatic disease.
* Metastases involving more than 6 liver segments.
* Radiographic evidence of involvement of the hepatic artery, major bile ducts, main portal vein, celiac/para aortic lymph nodes.
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2022-06-24 (Actual); Study Completion 2022-06-24 (Actual)

PRIMARY OUTCOMES:
Magnetic Resonance Displacement Encoding with Stimulated Echo (MR DENSE) imaging data of patients treated with chemotherapy prior to resection of metastases to explore its utility in detecting sinusoidal liver injury. | through study completion, an average of a year.

CONTACTS AND LOCATIONS:
Overall Officials: Priya Bhosale, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: M D Anderson Cancer Center — http://mdanderson.org